CLINICAL TRIAL: NCT03195452
Title: QD Isentress as Switch Strategy in Virologically Suppressed HIV-1 Infected-Patient
Brief Title: QDISS Stud: QD Isentress as Switch Strategy in Virologically Suppressed HIV-1 Infected-Patient
Acronym: QDISS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC16_0317
Record Dates: First submitted 2017-05-29; First posted 2017-06-22 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Virus-HIV
Keywords: HIV; Antiretrovirals; Raltegravir
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium

STUDY DESIGN:
Masking Description: Open label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Raltegravir (Experimental): antiretroviral tritherapy: Raltegravir 600 mg tablet orally (2 tablets QD) and 2 Nucleoside/Nucleotide reverse transcriptase inhibitor (NRTI)
  Interventions: Drug: Raltegravir and 2 Nucleoside/Nucleotide reverse transcriptase inhibitor (NRTI)

INTERVENTIONS:
Drug: Raltegravir and 2 Nucleoside/Nucleotide reverse transcriptase inhibitor (NRTI) — All virologically suppressed

SUMMARY:
Raltegravir (RAL) is a very effective antiretroviral drug with a favorable long term tolerability. RAL offers many advantages such as lack of drug-drug interactions, a good safety profile particularly on lipids, inflammation and bone parameters. Ral can be an very interesting for patient with comorbidities and comedications, intolerance or toxicities with their current ARV treatment. However its current formulation of one tablet of 400mg twice a day coul not suit many patients.

A new once-a-day formulation of RAL has been developed, with two tablets of 600 mg QD. Pharmacokinetic study in healthy volunteers has shown that this dosing provides increased RAL exposure compared to the standard formulation of 400 mg given twice a day.

The objective of this study is to evaluate the maintain of virologic suppression with raltegravir 600mg 2 tablets qd as part of a triple antiretroviral regimen in virologically controlled patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults of both gender ≥ 18 years
* Signed informed consent form
* Documented HIV-1 infection
* Stable antiretroviral therapy for ≥ 6 months consisting of 2 NRTIs (TDF/FTC or ABC/3TC )+ a 3rd agent either as a once or twice daily regimen, unless there is intolerance requiring change of therapy. In this situation of intolerance, patient with less than 6 months of current antiretroviral therapy will be allowed in the study.

As soon as TAF/FTC will be available in France, patients receiving TAF/FTC + 3rd agent could be enrolled.

Switch of TDF/FTC to TAF/FTC will be authorized as long as the change has occurred for more than 3 months prior to the screening visit. Such switch will be also allowed during the study, and, unless urgently needed, after the W24 visit.

Patients on stable raltegravir 400 mg 1 tablet twice daily plus 2 NRTI can be enrolled; number of these patients will be limited to 33% of the total cohort.

* Indication to current change antiretroviral therapy for at least one of the following reasons :

  1. Intolerance or prevention of toxicity
  2. Presence of a comorbid condition justifying change of the 3rd agent
  3. Management of drug-drug-interaction
  4. Patient's request, including switch to simplify or to improve convenience
* No prior virological failure on integrase-containing antiretroviral therapy or NNRTI-containing antiretroviral therapy or NRTI only-therapy
* HIV-1 RNA < 50 c/mL for ≥ 6 months. However, a single HIV-1 RNA ≥ 50 copies/mL and < 200 copies/mL with a subsequent HIV-1 RNA < 50 c/mL in the past 6 months is allowed.
* AST and ALT < 5 times the upper limit of normal
* Estimated glomerular filtration rate by MDRD equation >= 50 mL/min
* Hemoglobin > 8 g/dL
* Platelet count > 50 0000/mm3
* For women of childbearing potential: negative serum test for pregnancy and acceptance to use contraceptive methods
* Affiliation to a French Social Security program.

Exclusion Criteria:

* HIV-2 co-infection
* Concomitant treatments contra-indicated with raltegravir
* Patients receiving raltegravir 400mg, 2 tablets in one daily intake
* Patients with prior virological failure on NRTI+PI/r based regimen can be enrolled as long as historical plasma genotype and/or screening DNA genotype demonstrate absence of resistance or possible resistance to any drug. Subjects with previous failure to any other antiretroviral regimen cannot be enrolled.
* Presence of possible resistance or resistance to any nucleoside reverse transcriptase inhibitor or integrase inhibitor on a historical plasma genotype.
* Presence of possible resistance or resistance to any non- nucleoside reverse transcriptase inhibitor on a historical plasma genotype, with the exception of polymorphic mutations E138A/G/K/Q/R/S and V179D in patients naïve to NNRTI.
* Presence of resistance to any PI on a historical plasma genotype

In case were historical plasma genotype being not available or incomplete, resistance genotype will be performed on DNA at screening visit. Full treatment and cumulative resistance genotype history will have to be provided, at screening, to the principal investigator to approve any inclusion.

* For HCV co-infected patients, if specific treatment for hepatitis is required during the trial duration, such HCV therapy should be compatible with the ARV combination and only started after the W24 visit.
* HBV infection, in the absence of treatment with TDF or TAF
* Severe associated diseases requiring specific treatment, such as curative treatment of acute opportunistic infection
* Treatment with interferon, interleukin or any immunotherapeutic agent or chemotherapy
* Cancer diagnosis in the past 3 years with the exception of Kaposi sarcoma
* Subjects participating in another clinical trial evaluating therapies and having an exclusion period that is still ongoing during the screening phase
* Any condition which might compromise the safety of treatment and/or patient's adherence to trial procedures
* Person under guardianship, trusteeship or deprived of freedom by a judicial or administrative decision
* Difficulty in terms of follow-up (vacation, job transfer, geographical distance, lack of motivation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-05-06 (Actual)

PRIMARY OUTCOMES:
Number of copie/ml plasma HIV - RNA | 48 weeks

SECONDARY OUTCOMES:
Score evaluation of patient satisfaction | 48 weeks
Score evaluation of patient quality of life with PROQOL-HIV questionnaires | 48 weeks
Score evaluation of adherence | 48 weeks
Number of incidence of Treatment-Emergent Adverse Events | 48 weeks
Number of patient who have a viral load < 50 copies/ml | 48 weeks
number of discontinuation of Raltegravir | 48 weeks
number of treatment failure | 48 weeks
number of genotype resistance mutations | 48 weeks

CONTACTS AND LOCATIONS:
Locations (17):
- France (17):
  - CHU De Bordeaux, Bordeaux
  - CH de la Roche Sur Yon, La Roche-sur-Yon
  - CH du Mans, Le Mans
  - CHU de Lyon, Lyon
  - CHRU de Montpellier, Montpellier
  - CHU of NANTES, Nantes
  - CHU de Nice, Nice
  - CHR orléans, Orléans
  - CHU de Bichat, Paris
  - CHu hotel dieu, Paris
  - CHU la pitié, Paris
  - Hopital Avicenne, Paris
  - Hopital Necker, Paris
  - Hopital St Louis, Paris
  - CHU de Reims, Reims
  - CH de Tourcoing, Tourcoing
  - CHRU de Tours, Tours

REFERENCES:
- [Derived] Hall N, Allavena C, Katlama C, Jobert A, Molina JM, Cua E, Bani-Sadr F, Hocqueloux L, Duvivier C, Merrien D, Hikombo H, Andre-Garnier E, Gaultier A, Raffi F; QDISS Study Group. Raltegravir 1200 mg once daily as maintenance therapy in virologically suppressed HIV-1 infected adults: QDISS open-label trial. AIDS Res Ther. 2022 Jan 15;19(1):4. doi: 10.1186/s12981-022-00428-5. PMID 35033092